CLINICAL TRIAL: NCT01972074
Title: Behavioral and Neural Response to Memantine in Adolescents With Autism Spectrum Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Assistant Professor of Psychiatry, Harvard Medical School; Medical Director, Bressler Program for Autism Spectrum Disorder, Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-P-001826
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Treatment; Adolescents; Memantine; functional Magnetic Resonance Imaging; MRS; Neuroimaging
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Memantine (Experimental): Participants in the placebo arm will receive placebo (no active ingredients) in capsule form twice daily. It will be administered twice daily for 12 weeks. Participants will undergo neuroimaging before and after the 12-week treatment phase.
  Placebo: Capsule
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Participants in the memantine arm will receive memantine in capsule form twice daily. It will be administered twice daily for 12 weeks (including a 4-week titration phase to a maximum dose of 20 mg per day). Participants will undergo neuroimaging before and after the 12-week treatment phase.
  Memantine: Capsule
  Interventions: Other: Placebo
- Control Group (No Intervention): Healthy controls will undergo neuroimaging twice (12 weeks apart) and will receive no intervention during the 12-week window.

INTERVENTIONS:
Drug: Memantine — Capsule
  Other Names: Namenda
  Arms: Memantine
Other: Placebo — Capsule
  Arms: Placebo

SUMMARY:
This study is a 12-week, randomized-controlled trial of memantine hydrochloride (Namenda) for the treatment of social impairment in adolescents with autism spectrum disorder (ASD). The investigators will also conduct pre- and post-treatment neuroimaging (functional magnetic resonance imaging [fMRI] and hydrogen magnetic resonance spectroscopy [HMRS]) to assess neural functional deficits in adolescents with autism spectrum disorder compared to healthy volunteer adolescents. This pre- and post-neuroimaging will also be used to assess any effects of memantine therapy on neural function in adolescents with autism spectrum disorder. The investigators hypothesize that short-term memantine monotherapy will be safe, well-tolerated, and effective in improving the core symptoms of autism spectrum disorder in adolescents with autism spectrum disorder. Additionally, the investigators hypothesize that following memantine therapy, adolescents with autism spectrum disorder will exhibit a decrease in glutamate (Glu) concentration in the anterior cingulate cortex (ACC) and a change towards normalization in altered functional connectivity of the anterior cingulate cortex and medial temporal lobes, consistent with improvement in social impairments in autism spectrum disorder. The investigators hypothesize that compared to healthy volunteer participants, participants with autism spectrum disorder will significantly differ on neuroimaging measures at baseline but that following memantine therapy, the difference between autism spectrum disorder and healthy volunteer neuroimaging data will decrease.

ELIGIBILITY:
INCLUSION CRITERIA

All Participants:

1. Male and female participants, ages 8-17 years (inclusive)

   Participants with Autism Spectrum Disorder:
2. Meets Diagnostic and Statistical Manual-5 autism spectrum disorder diagnostic criteria, as established by clinical diagnostic interview
3. At least moderate severity of social impairment, as measured by a total raw score of ≥85 on the parent/guardian-completed Social Responsiveness Scale, Second Edition (SRS-2) and a score of ≥4 on the clinician-administered Autism Spectrum Disorder Clinical Global Impression-Severity scale (ASD CGI-S)

Healthy Control Participants:

2. Age-, sex-, and IQ-matched with participants with autism spectrum disorder 3. No Axis I diagnoses, as established by the Kiddie Schedule for Affective Disorders and Schizophrenia-Epidemiological Version (K-SADS-E) and confirmed by clinical diagnostic interview 4. No significant traits of autism spectrum disorder, as measured by a total raw score of <60 on the parent/guardian-completed Social Responsiveness Scale, Second Edition

EXCLUSION CRITERIA

All Participants:

1. IQ ≤70 based, on the Wechsler Abbreviated Scale of Intelligence, Second Edition (WASI-II) Vocabulary and Matrix Reasoning subtests
2. Impaired communicative speech
3. Current treatment with the following medications, which are known to impact glutamate levels:

   1. Lamotrigine
   2. Amantadine
   3. N-acetylcysteine
   4. D-cycloserine
4. Current treatment with a psychotropic medication, not listed above, on a dose that has not been stable for at least 4 weeks prior to study baseline
5. Co-administration of drugs that compete with memantine for renal elimination using the same renal cationic system, including hydrochlorothiazide, triamterene, metformin, cimetidine, ranitidine, quinidine, and nicotine
6. Initiation of a new psychosocial intervention within 30 days prior to randomization
7. Participants who are pregnant and/or nursing
8. Participants with a history of non-febrile seizures without a clear and resolved etiology
9. Participants with a history of or a current liver or kidney disease
10. Clinically unstable psychiatric conditions or judged to be at serious suicidal risk
11. Participants who meet for alcohol or drug dependence or abuse on the Kiddie Schedule for Affective Disorders and Schizophrenia-Epidemiological Version. If the participant has a recent history of substance abuse, as an added precaution, there will be a 2-week washout period before initiating the trial. There are no known safety issues relating to memantine and recent history of substance abuse.
12. Serious, stable or unstable, systemic illness, including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease
13. Participants with severe hepatic impairment (Liver Function Tests [LFTs] >3 times the Upper Limit of Normal [ULN])
14. Participants with genitourinary conditions that raise urine Power of Hydrogen (pH) (e.g., renal tubular acidosis, severe infection of the urinary tract)
15. Known hypersensitivity to memantine
16. Severe allergies or multiple adverse drug reactions
17. A non-responder or history of intolerance to memantine after treatment at adequate doses, as determined by the clinician
18. Investigator and his/her immediate family, defined as the Investigator's spouse, parent, child, grandparent, or grandchild.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Joshi G, Gonenc A, DiSalvo M, Faraone SV, Ceranoglu TA, Yule AM, Uchida M, McDougle CJ, Wozniak J. Memantine to Treat Social Impairment in Youths With Autism Spectrum Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2534927. doi: 10.1001/jamanetworkopen.2025.34927. PMID 41032298
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Brignell A, Marraffa C, Williams K, May T. Memantine for autism spectrum disorder. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013845. doi: 10.1002/14651858.CD013845.pub2. PMID 36006807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited for 3 years (2015 - 2018). They were recruited from existing and new patients at 3 Massachusetts General Hospital sites: Bressler Program for Autism Spectrum Disorder, Lurie Center for Autism, and Child and Adolescent Outpatient Psychiatry Clinic. Participants were also recruited using flyers and internet advertisements.
Pre-assignment Details: Per protocol, participants were enrolled when they provided informed consent. They then underwent screening procedures to confirm eligibility. If eligible and willing/able to participate, participants then began study procedures. Some participants dropped out prior to starting study procedures and were, therefore, excluded from this analysis.
Groups:
- Memantine: Participants in the memantine arm will receive memantine in capsule form twice daily. It will be administered twice daily for 12 weeks (including a 4-week titration phase to a maximum dose of 20 mg per day). Participants will undergo neuroimaging before and after the 12-week treatment phase.
  Memantine: Capsule
- Placebo: Participants in the placebo arm will receive placebo (no active ingredients) in capsule form twice daily. It will be administered twice daily for 12 weeks. Participants will undergo neuroimaging before and after the 12-week treatment phase.
  Placebo: Capsule
Period: Overall Study
Arm/Group | Memantine | Placebo | Control Group
Started | 22 | 21 | 18
Completed | 16 | 17 | 15
Not Completed | 6 | 4 | 3
Not completed — Adverse Event | 4 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Scanner Unavailable | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Participants in the Memantine and Placebo groups completed the Week 0: Baseline study visit. Baseline Participants in the Control group completed the Week 100: Baseline Scan study visit. The Baseline assignment is different for the Control group because they received no intervention and so did not complete the Week 0: Baseline study visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Control Group | Total
Number analyzed (Participants) | 22 | 21 | 18 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 21 | 18 | 61
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (2.7) | 13.3 (2.5) | 12.6 (2.7) | 13.0 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 16
  Male | 17 | 16 | 12 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 21 | 20 | 17 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 20 | 15 | 55
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 18 | 61

OUTCOME MEASURES:

1. Primary Outcome: Treatment Responder
Description: Treatment responders are defined as having a 25% reduction, from baseline to endpoint, in Social Responsiveness Scale, Second Edition: School-Age, Parent Report (SRS-2) total raw score and an Autism Spectrum Disorder Clinical Global Impression-Improvement (ASD CGI-I) score ≤2. The Social Responsiveness Scale, Second Edition (SRS-2) is a 65-item rating scale completed by the parents/guardians of children ages 4-18. It is used to measure the severity of autism spectrum disorder symptoms. Each item is rated on a 4-point Likert scale, ranging from 1=Not True to 4=Almost Always True. Higher scores indicate a higher severity of autism spectrum disorder symptoms. The Autism Spectrum Disorder Clinical Global Impression-Improvement subscale (ASD CGI-I) is a clinician-rated measure of the improvement of autism spectrum disorder symptoms. The subscale is rated on a 7-point Likert scale, ranging from 1=Very Much Improved to 7=Very Much Worse. Higher scores indicate less symptom improvement.
Time Frame: 12 Weeks (from Baseline [Week 0] to Endpoint [Week 12])
Population: Participants included in this analysis were exposed to study medication for at least 2 weeks. Participants in the Control Group were excluded from this analysis because they did not receive study medication and, therefore, cannot be categorized into Treatment Responders vs. Treatment Non-Responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 19 | 21
Participants | 9 | 4

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Adverse events were collected from participants in the memantine arm and the placebo arm systematically, via regular investigator assessment. At every study visit, study clinicians queried participants and their parent(s)/guardian(s) about any adverse events that may have occurred since the last study visit. Participants in the Control Group were excluded from this analysis because they did not receive study medication and adverse events were not monitored/assessed for the Control Group.
Arm/Group | Memantine | Placebo | Control Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/0
Other Adverse Events (participants affected / at risk) | 14/22 | 9/21 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=22) | Placebo (N=21) | Control Group (N=0)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Anxious/Worried (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Cold/Infection/Allergy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizzy/Lightheaded (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 2 (2) | 0 (0)
Increased Appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Increased Bed Wetting (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Irritability & Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Self-Harm (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT01972074/Prot_SAP_000.pdf